CLINICAL TRIAL: NCT01453608
Title: A Randomised, Double-blind Controlled Phase 4 Study to Compare the Efficacy and Safety of Intravenous Ferric Carboxymaltose With Placebo in Patients With Chronic Heart Failure and Iron Deficiency
Brief Title: A Study to Compare the Use of Ferric Carboxymaltose With Placebo in Patients With Chronic Heart Failure and Iron Deficiency
Acronym: CONFIRM-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FER-CARS-05
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Iron Deficiency; Chronic Heart Failure
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferinject (ferric carboxymaltose) (Experimental)
  Interventions: Drug: Ferinject (ferric carboxymaltose)
- Placebo (saline) (Placebo Comparator)
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Drug: Ferinject (ferric carboxymaltose) — Subjects will receive Ferinject (ferric carboxymaltose) intravenously on Day 0
  Arms: Ferinject (ferric carboxymaltose)
Drug: Placebo (saline) — Subjects will receive Placebo (saline) intravenously on Day 0
  Arms: Placebo (saline)

SUMMARY:
The purpose of this study is to determine, relative to placebo, the effect of iron repletion therapy using intravenous (IV) ferric carboxymaltose on exercise capacity in patients with chronic heart failure and iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Iron deficient subjects with stable chronic heart failure (CHF) (NYHA II-III) on optimal background therapy for CHF
* Reduced left ventricular ejection fraction
* Capable of completing 6 minute walk test
* At least 18 years of age and with written informed consent prior to any study specific procedures

Exclusion Criteria:

* Erythropoietin stimulating agent (ESA) use, IV iron therapy and/or blood transfusion in previous 6 weeks prior to randomisation
* Exercise training program(s) in the 3 months prior to screening or planned in the next 6 months
* Chronic liver disease and/or elevated liver enzymes
* Vitamin B12 and/or serum folate deficiency
* Subject is not using adequate contraceptive precautions during the study
* Body weight ≤ 35 kg
* No other significant cardiac or general disorders that would compromise the ability to give informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in six minute walk test from baseline to week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, MD, Principal Investigator — Cardiology Department - Centre for Heart Disease - Clinical Military Hospital
Locations (2):
- Clinical Military Hospital, Wroclaw, Poland
- State Educational Institution of Higer Professional Education, Ryazan, Russia

REFERENCES:
- [Derived] Ponikowski P, van Veldhuisen DJ, Comin-Colet J, Ertl G, Komajda M, Mareev V, McDonagh T, Parkhomenko A, Tavazzi L, Levesque V, Mori C, Roubert B, Filippatos G, Ruschitzka F, Anker SD; CONFIRM-HF Investigators. Beneficial effects of long-term intravenous iron therapy with ferric carboxymaltose in patients with symptomatic heart failure and iron deficiencydagger. Eur Heart J. 2015 Mar 14;36(11):657-68. doi: 10.1093/eurheartj/ehu385. Epub 2014 Aug 31. PMID 25176939